CLINICAL TRIAL: NCT02217007
Title: A Phase 2a, Open-Label Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of Orally Administered SNC-102 in Subjects With Tourette Syndrome
Brief Title: A Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of SNC-102 in Subjects With Tourette Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding stopped, company closed
Sponsor: Synchroneuron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC-102-211 TS
Record Dates: First submitted 2014-07-23; First posted 2014-08-15 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Tourette Syndrome
Keywords: Tourette; Tourette's; tic
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNC-102 sustained release tablet (Experimental): SNC-102 oral tablet 4 weeks at 800mg BID plus 4 weeks at 1600mg in the morning and 800mg in the evening
  Interventions: Drug: SNC-102 sustained release tablet

INTERVENTIONS:
Drug: SNC-102 sustained release tablet — SNC-102 is an 800 mg tablet. It will be administered twice daily (morning and evening) for a total of 8 weeks: the initial 4 weeks will be 1 tablet in the morning and 1 tablet in the evening; the next 4 weeks will be 2 tablets in the morning and 1 tablet in the evening.
  Other Names: SNC-102; acamprosate calcium sustained release tablet; acamprosate calcium; acamprosate

SUMMARY:
This is an open-label study of SNC-102 (acamprosate calcium sustained release tablet) in adult subjects with Tourette Syndrome. Subjects will be treated with oral doses of SNC-102 800 mg on a BID basis - before breakfast and at bedtime - for 4 weeks and the same subjects will be treated with SNC-102 1600mg in the morning and 800mg in the evening for an additional 4 weeks. Subjects will be assessed for changes in tic severity, safety, and pharmacokinetics. The study hypothesis is that treatment with SNC-102 will improve the tic severity in adult subjects with Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by a Board-certified neurologist or psychiatrist of Tourette Syndrome according to Diagnostic and Statistical Manual (DSM)-V criteria for Tourette's Disorder, viz.
* Both multiple motor and one or more vocal tics have been present at some time during the illness, although not necessarily concurrently.
* The tics may wax and wane in frequency but have persisted for more than 1 year since first tic onset.
* Onset is before age 18 years.
* The disturbance is not attributable to the physiological effects of a substance (e.g., cocaine) or another medical condition (e.g., Huntington's disease, postviral encephalitis).
* Moderate to severe tics as indicated by a Clinical Global Impression (CGI) score of 4 or higher on both the Screening Visit and the Baseline Visit while on their usual drug therapy for Tourette Syndrome.
* If using a permitted medication (SSRI, Serotonin-norepinephrine reuptake inhibitors (SNRI), alpha-2 agonist, benzodiazepine, dopamine antagonist, or stimulant) the dose has been stable for at least 4 weeks prior to the Screening Visit and is expected to remain stable through the conclusion of the study.
* Ability to swallow investigational tablets whole and without chewing, as demonstrated by swallowing a placebo tablet at the Screening Visit.

Exclusion Criteria:

* Diagnosis of epilepsy.
* Treatment with an antiepileptic drug with the exception of a stable dose of clonazepam. Topiramate and lamotrigine are specifically excluded.
* Unstable psychiatric status, as indicated by any change in psychotropic medication (unless approved by the Sponsor), or by psychiatric hospitalization, within 30 days prior to the Screening Visit.
* Active drug or alcohol dependence or abuse.
* Current use of cocaine, amphetamine, phencyclidine, or ketamine, documented either by history or by urinary drug screening at Screening and Baseline Visits. Drugs used to treat attention deficit-hyperactivity disorder or obsessive-compulsive symptoms are allowed if stable for at least 4 weeks prior to the Screening Visit and are expected to remain stable through the course of the trial. Any other drugs identified on drug screening will warrant exclusion only if the Principal Investigator, in consultation with the Sponsor, judges that their presence could interfere with the objectives of the trial.
* Risk of significant medication non-adherence, based on the judgment of the Principal Investigator.
* History of neuroleptic malignant syndrome.
* Significant risk, in the judgment of the Principal Investigator, of suicidal or violent behavior.
* Female subjects with a history of pre-menstrual exacerbation of tics.
* Initiation of oral contraceptive medication, insertion of progestin contraceptive implant, or change in dose, within 30 days prior to the Screening Visit, or anticipated while participating in the trial.
* History of short-bowel or other malabsorption syndrome, gastrointestinal hypermotility of any cause, or any gastrointestinal disease or surgery that, in the judgment of the Principal Investigator, could interfere with absorption of orally-administered medication, reduce intestinal transit time or pre-dispose to gastric outlet obstruction.
* Allergy or intolerance to acamprosate.
* Prior treatment with acamprosate for any indication.
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
* Use of any investigational agents within 4 weeks of Baseline.
* Pregnant or lactating female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in total tic severity score on the Yale Global Tic Severity Scale at 4 weeks | 4 weeks
  Determine whether SNC-102 800 mg twice daily (BID) will decrease tic severity in adult patients with Tourette Syndrome (TS), as measured by changes from baseline to 4 weeks in the total tic severity score on the Yale Global Tic Severity Scale (Y-GTSS).
Improvement in total tic severity score on the Yale Global Tic Severity Scale at 8 weeks | 8 weeks
  Determine whether SNC-102 1600 mg in the morning and 800 mg in the evening will decrease tic severity in adult patients with Tourette Syndrome (TS) as measured by change from baseline to Day 57 in the total tic severity score on the Yale Global Tic Severity Scale (Y-GTSS).

SECONDARY OUTCOMES:
Assess safety and tolerability | 2, 4, 6, 8, 11 weeks
  Assess the safety and tolerability of SNC-102 in the adult TS population, including assessing the effects, if any, of SNC-102 on symptoms of depression, anxiety, obsessive-compulsive disorder (OCD), and attention deficit-hyperactivity disorder (ADHD);
Evaluate clinical effects of SNC-102 on tic severity at 2 weeks and 6 weeks | 2, 6 weeks
  Further evaluate the clinical effects of SNC-102 in this population as measured by changes from baseline in Y-GTSS total tic severity score at 2 weeks and 6 weeks
Pharmacokinetic profile of SNC-102 in Tourette Syndrome subjects | 2, 4, 6, 8 weeks
  Assess the pharmacokinetics (PK) of acamprosate administered as SNC-102, including measures of the plasma concentration at 3 hours post-dose (C3h) and the trough plasma concentration (Cmin). The pharmacokinetic analysis will be based on the pre-dose and 3 hour post-dose plasma concentrations of acamprosate on the first day of dosing (Baseline) and on the Day 15, Day 29, Day 43 and Day 57 visits.
Explore relationship between study drug plasma levels and the magnitude of clinical response | 2, 4, 6, 8 weeks
  Explore the relationship between steady-state acamprosate plasma levels and the magnitude of clinical response to the drug.
Evaluate clinical effects of SNC-102 on Global Clinical Impression | 2, 4, 6, 8, 11 weeks
  Evaluate the clinical effects of SNC-102 in this population as measured by changes from baseline in Clinical Global Impression (CGI) at all post-baseline visits
Evaluate clinical effects of SNC-102 on tic severity sub scales | 2, 4, 6, 8, 11 weeks
  Further evaluate the clinical effects of SNC-102 in this population as measured by changes from baseline in Y-GTSS sub scales at all visits

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Fogel, MD, Study Director — Synchroneuron Inc.
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - North Shore University Hospital, Dept. of Psychiatry, Manhasset, New York